CLINICAL TRIAL: NCT05367323
Title: Is Pain Pressure Threshold Consistent With the Biomechanical-Viscoelastic Changes for L4-5 Supraspinous Ligament in Women Undergoing Midline Spinal Anaesthesia for Cesarean Delivery
Brief Title: Pain Pressure Threshold Values Versus the Biomechanical-Viscoelastic Findings of L4-5 Supraspinous Ligament in Women Who Underwent Cesarean Delivery With Spinal Anaesthesia
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Assistant Lecturer of Physical Therapy for Women's Health, South Valley University
Other Study IDs: Algometry VS Myoton PRO
Record Dates: First submitted 2022-04-27; First posted 2022-05-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Low Back Biomechanical Dysfunctions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: 22 women who underwent cesarean delivery using spinal anesthesia
  Interventions: Device: Pressure algometry (Baseline 2.2-Pound Dolorimeter) and Myoton PRO device (MyotonPRO; Myoton AS, Tallinn, Estonia)
- Group B: 22 women who were in the control group (they never experience pregnancy, or anaesthesia)
  Interventions: Device: Pressure algometry (Baseline 2.2-Pound Dolorimeter) and Myoton PRO device (MyotonPRO; Myoton AS, Tallinn, Estonia)

INTERVENTIONS:
Device: Pressure algometry (Baseline 2.2-Pound Dolorimeter) and Myoton PRO device (MyotonPRO; Myoton AS, Tallinn, Estonia) — Both instruments are used for the assessment of the L4-5 interspinous space pain pressure threshold and the biomechanical-viscoelastic properties of L4-5 supraspinous ligament respectively
  Other Names: Myoton PRO device (MyotonPRO; Myoton AS, Tallinn, Estonia)

SUMMARY:
Cesarean delivery is a major obstetric surgery that aims to save the lives of mothers and their neonates from complications that may be related to high-risk pregnancy and difficult delivery (Teguete et al., 2012). According to the updated Egyptian demographic and health survey, the rate of cesarean delivery in Egypt has increased until it reached about 52 % of all deliveries (Abdel-Tawab et al., 2018).

Neuraxial anesthesia, especially spinal anaesthesia has been and continues to be the gold standard anesthesia for cesarean section (Mhyre and Sultan., 2019).

DETAILED DESCRIPTION:
Low back pain (LBP) after neuraxial anaesthesia is a typical mild intensity pain. It is thought to be caused by needle trauma and local anaesthetic myotoxicity. Post-dural puncture backache (PDPB), which is defined as a persistent pain around the puncture site without radicular pain, is a common consequence following spinal anaesthesia (Benzon et al., 2016). Back pain following anaesthesia may be attributed to ligament, fascia, or bone injuries with localized bleeding; rigidity of the spine; anaesthesia-induced relaxation of the paraspinal muscles; flattening of the typical lumbar convexity, and stretching and straining of the lumbosacral ligaments and joint capsules (Benzon et al., 2016).

Pressure algometry is an objective well-known and well-validated method which induces acute experimental pain for determining the Pain Pressure Threshold (PPT) in various parts of the body (Pelfort et al., 2015). The PPT is a quantitative sensory value for tissue sensitivity that is defined as the smallest amount of pressure that causes pain (Ylinen., 2007).

The MyotonPRO is a portable valid device for measuring the biomechanical properties such as stiffness and the viscoelasticity of the superficial myofascial tissue objectively (Nguyen et al., 2022). Stiffness, stress relaxation time and creep are biomechanical and viscoelastic properties of lower lumbar myofascia that can be measured using the MyotonPRO device either in healthy adults or low back pain patients (Ilahi et al., 2020). Also, the MyotonPRO can tell the difference between a trigger point and a non-trigger point in terms of viscoelastic qualities such as stress relaxation time or creeping through objective assessment (Roch et al., 2020).

Stiffness is defined as a biomechanical property that represents the resistance to deformation which is directly related to the clinical measurement of muscle tone felt during palpation (Nordin andFrankel., 2012). Both stress relaxation time and creep are viscoelastic properties of the myofascia. Stress relaxation time means the time for a muscle to return to its original shape from deformation after the removal of the causative external load. However, Creep is defined as the gradual lengthening of a muscle and connective tissues over time when put under persistent tensile stress (Myoton., 2013).

In this study we will investigate if the midline spinal anaesthesia for cesarean delivery will be associated with decreased L4-5 interspinous pain pressure threshold - lower PPT yields higher pain - after cesarean delivery or not, and we will compare these findings of L4-5 interspinous pain pressure threshold and the biomechanical properties (stiffness, relaxation time and creeping) of L4-5 supraspinous ligament. Due to the lack of previous objective studies and to fill the gap in this point, this study will be considered the first conducted study to answer our research question.

The null hypothesis indicates that spinal anaesthesia for cesarean delivery has neither a relative risk for decreased L4-5 interspinous pain pressure threshold nor L4-5 supraspinous ligament biomechanical changes.

ELIGIBILITY:
Inclusion Criteria:

1. All women in the epidural and spinal anesthetic groups gave birth through a cesarean delivery.
2. All women either primiparous or multiparous have not had anesthesia (epidural, spinal ) for at least one year prior to the last obstetric anesthesia.
3. Their ages ranged from 18 to 35 years.
4. All participants had a body mass index (BMI), of not more than 30, and a waist to hip ratio of not more than 1.
5. Participants were assessed between the 6th week to the 12th week postnatal.
6. All participants were able to continue all assessment procedures.
7. They were medically stable.

Exclusion Criteria:

1. Women who delivered through vaginal delivery.
2. Women who delivered through cesarean delivery, but the used anesthetic technique was the paramedian approach of spinal anesthesia.
3. Women with urinary tract infections and diastasis recti.
4. Women who were below 18 years old or above 35 years old.
5. Women who had (BMI) above 30 or waist to hip ratio above 1.
6. Women who did not continue all assessment procedures.
7. Women who had any non-myofascial low back dysfunctions as women who were diagnosed with lumbar disc prolapse or spondylolisthesis.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — All participants were females as this study related to the Department of Physical Therapy for Women's Health
Study Population: Retrospective Cohort Study in which 44 women participated in this study. They were selected from South Valley University Teaching Hospitals.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
L4-5 Supraspinous Ligament Pain pressure threshold in Pounds | Assessment will be done 6-12 weeks after the use of anaesthesia during Cesarean section
  The PPT is a quantitative sensory value for tissue sensitivity that is defined as the smallest amount of pressure that causes pain

SECONDARY OUTCOMES:
L4-5 supraspinous ligament Stiffness in Newton/meter | Assessment will be done 6-12 weeks after the use of anaesthesia during Cesarean section
  The MyotonPRO device measures Stiffness which is defined as a biomechanical property that represent the resistance to deformation which is directly related to the clinical measurement of muscle tone felt during palpation
L4-5 supraspinous ligament Stress Relaxation Time in milliseconds | Assessment will be done 6-12 weeks after the use of anaesthesia during Cesarean section
  The MyotonPRO device measures Stress relaxation time which means the time for a muscle to return to its original shape from deformation after removal of the causative external load
L4-5 supraspinous ligament Creep in Deborah number | Assessment will be done 6-12 weeks after the use of anaesthesia during Cesarean section
  The MyotonPRO device measures Creep that is defined as the gradual lengthening of a muscle and connective tissues over time when put under a persistent tensile stress

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, South Valley University, Qina, Qena Governorate, Egypt